CLINICAL TRIAL: NCT06375421
Title: Development of Ecological Momentary Intervention for Memory in Chronic Traumatic Brain Injury: A Pilot and Feasibility Study
Brief Title: Pilot and Feasibility of MEMI for Chronic Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Emily Morrow, Postdoctoral Research Fellow, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: GR018280
Record Dates: First submitted 2024-04-08; First posted 2024-04-19 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; memory; ecological momentary intervention
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: The order of conditions and the order of word list presentation will be counterbalanced. The order of condition/word list combination will be pre-determined, and participants will be assigned to the next available combination based on when they join the study (i.e., a counterbalanced within-person crossover design).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention, then Active Comparator (Other): Participants complete the Intervention (MEMI spaced retrieval) week, followed by the Active Comparator (blocked retrieval) week.
  Interventions: Behavioral: MEMI (Memory Ecological Momentary Intervention) Spaced Retrieval; Behavioral: Blocked Retrieval
- Active Comparator, then Intervention (Other): Participants complete the Active Comparator (blocked retrieval) week, followed by the Intervention (MEMI spaced retrieval) week.
  Interventions: Behavioral: MEMI (Memory Ecological Momentary Intervention) Spaced Retrieval; Behavioral: Blocked Retrieval

INTERVENTIONS:
Behavioral: MEMI (Memory Ecological Momentary Intervention) Spaced Retrieval — Participants complete their initial learning session, and the subsequent retrieval sessions are spaced out over the course of the week (two short retrieval sessions each day) using MEMI. Then, they complete a 15-minute test for their memory of all of the trained items at the end of the week.
Behavioral: Blocked Retrieval — Participants will complete their initial learning session on the target words, then immediately receive all of the exposures to each of the items in a single block. They do not complete any more retrieval sessions until one week later, when they complete a 15-minute test for their memory of all of the trained items.

SUMMARY:
This is a pilot and feasibility study for a mobile phone-delivered intervention for memory, called MEMI (memory ecological momentary intervention), that was designed to support adults with chronic traumatic brain injury with their memory. The goal of the study is to examine the feasibility and acceptability of MEMI and to assess preliminary efficacy as to whether technology-delivered spaced memory retrieval opportunities improve memory in people with and without a history of chronic traumatic brain injury.

DETAILED DESCRIPTION:
Deficits in memory and learning are hallmark to traumatic brain injury (TBI) and limit a person's ability to participate in medical care, benefit from therapy, maintain positive social relationships, and be successful at school or work. There has been limited progress in the last several decades in advancing functional memory outcomes after TBI, and constraints in the timing and context of the existing rehabilitation model may contribute. In memory rehabilitation, each opportunity to retrieve information strengthens that information in the neocortex, and is thus both an assessment and a learning opportunity. Increasing the contextual diversity of learning opportunities (i.e., in the daily lives and contexts of patients) may improve the rehabilitation potential of patients with TBI.

This study is a pilot and feasibility trial of MEMI as a technology-delivered intervention that extends memory assessment and treatment over time and space. We use a counterbalanced within-participant crossover design to examine MEMI's feasibility and acceptability in daily life and collect preliminary efficacy data as to how using MEMI in daily life affects long-term recall for participants with and without TBI. The study includes a group of adults with a chronic history of moderate-severe TBI and a demographically matched control group. Each participant uses MEMI for two weeks, each in a different condition:

* Blocked (Active Comparator) Condition: During one of the weeks, participants will complete their initial learning session on the target words, then immediately receive all of the exposures to each of the items in a single block. They do not complete any more retrieval sessions until one week later, when they complete a 15-minute test for their memory of all of the trained items.
* Spaced (MEMI Intervention) Condition: During the other week, participants complete their initial learning session, and the subsequent retrieval sessions are spaced out over the course of the week (two short retrieval sessions each day) using MEMI. Then, they complete a 15-minute test for their memory of all of the trained items at the end of the week.

This study addresses three aims:

Aim 1: To examine the real-world feasibility and acceptability of MEMI via user engagement and survey data.

Aim 2: To explore preliminary efficacy of spaced retrieval via MEMI to improve long-term word recall in individuals with and without chronic TBI.

Aim 3: To explore how a) spatial context and b) temporal context of exposures affect long- term word recall in people with and without chronic TBI.

ELIGIBILITY:
Inclusion criteria:

For participants with TBI:

* Moderate-severe TBI. All participants were determined to have a history of moderate-severe TBI upon joining the Vanderbilt Brain Injury Patient Registry. This determination was made based on the Mayo Classification Scale.
* All participants are at least 6 months post-injury at the time of study enrollment and thus exhibit chronic and stable neuropsychological profiles.
* Age ranging from 18-60, to rule out developmental TBI and limit influence of age-related cognitive decline.

For all participants:

* Oral and written language skills sufficient for the study tasks. This will be screened in the initial video conference contact with the participant, when consent is obtained.
* Participants must own a smartphone to access the Gorilla online behavioral experiment platform from their mobile phones.

Exclusion criteria:

For participants with TBI:

• History of medical or neurological disease affecting the brain or language, before or after the qualifying TBI.

For non-injured comparison peers:

• History of neurological or cognitive disability, including TBI

For all participants:

* Any disability (e.g., vision impairment, hard of hearing, aphasia or other neurologic condition) that limits ability to read, type, or verbally communicate.
* Demonstrates inability to receive and respond to a text message after training by study personnel.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Morrow, Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the pilot trial will be de-identified and made available following publication of the results to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months after results publication. No end date.
Access Criteria: Approval of a proposal by the study PI.

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Traumatic Brain Injury (TBI): Intervention, Then Active Comparator; Non-Injured Comparison Participants: Intervention, Then Active Comparator: Participants complete the Intervention (MEMI spaced retrieval) week, followed by the Active Comparator (blocked retrieval) week.
- Participants With Traumatic Brain Injury (TBI): Active Comparator, Then Intervention; Non-injured Comparison Participants: Active Comparator, Then Intervention: Participants complete the Active Comparator (blocked retrieval) week, followed by the Intervention (MEMI spaced retrieval) week.
Period: First Intervention (1 Week)
Arm/Group | Participants With Traumatic Brain Injury (TBI): Intervention, Then Active Comparator | Non-Injured Comparison Participants: Intervention, Then Active Comparator | Participants With Traumatic Brain Injury (TBI): Active Comparator, Then Intervention | Non-injured Comparison Participants: Active Comparator, Then Intervention
Started | 10 | 10 | 10 | 10
Completed | 9 | 10 | 9 | 10
Not Completed | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Period: Second Intervention (1 Week)
Arm/Group | Participants With Traumatic Brain Injury (TBI): Intervention, Then Active Comparator | Non-Injured Comparison Participants: Intervention, Then Active Comparator | Participants With Traumatic Brain Injury (TBI): Active Comparator, Then Intervention | Non-injured Comparison Participants: Active Comparator, Then Intervention
Started | 9 | 10 | 9 | 10
Completed | 9 | 10 | 9 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants With Traumatic Brain Injury (TBI): Participants with TBI were in the chronic phrase (>6 months post-injury). TBI severity was moderate-severe per the Mayo Classification System. Participants were 18-55 years of age to exclude developmental effects of TBI and conservatively limit the effects of age-related cognitive decline. Participants with TBI had no other neurological or cognitive disabilities aside from the qualifying injury.
- Non-injured Comparison Participants: Comparison participants were also 18-55 years of age, had no history of neurological or cognitive disability, and were matched to the participants with TBI on age, sex, and education.
- Total: Total of all reporting groups
Arm/Group | Participants With Traumatic Brain Injury (TBI) | Non-injured Comparison Participants | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (10.4) | 40.7 (9.8) | 40.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 19 | 19
  Not Hispanic or Latino | 20 | 1 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 20 | 16 | 36
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Educational Attainment [Mean (Standard Deviation); unit: years] | 14.7 (2.3) | 14.6 (2.3) | 14.6 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability
Description: Acceptability of Intervention Measure (4 = completely disagree/not acceptable - worse, 20 = completely agree/acceptable - better)
Time Frame: 1 week in each intervention condition
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Participants With Traumatic Brain Injury (TBI) Completing Intervention (MEMI Spaced Retrieval); Non-Injured Comparison Participants Completing Intervention (MEMI Spaced Retrieval): MEMI (Memory Ecological Momentary Intervention) Spaced Retrieval: Participants complete their initial learning session, and the subsequent retrieval sessions are spaced out over the course of the week (two short retrieval sessions each day) using MEMI. Then, they complete a 15-minute test for their memory of all of the trained items at the end of the week.
- Participants With Traumatic Brain Injury (TBI) Completing Active Comparator (Blocked Retrieval); Non-injured Comparison Participants Completing Active Comparator (Blocked Retrieval): Blocked Retrieval: Participants will complete their initial learning session on the target words, then immediately receive all of the exposures to each of the items in a single block. They do not complete any more retrieval sessions until one week later, when they complete a 15-minute test for their memory of all of the trained items.
Arm/Group | Participants With Traumatic Brain Injury (TBI) Completing Intervention (MEMI Spaced Retrieval) | Non-Injured Comparison Participants Completing Intervention (MEMI Spaced Retrieval) | Participants With Traumatic Brain Injury (TBI) Completing Active Comparator (Blocked Retrieval) | Non-injured Comparison Participants Completing Active Comparator (Blocked Retrieval)
Number analyzed (Participants) | 19 | 20 | 19 | 20
score on a scale | 16.68 (2.81) | 17.55 (2.18) | 15.31 (4.50) | 17.25 (2.79)

2. Primary Outcome: Feasibility (Engagement)
Description: Number of possible sessions that participants complete in each condition (min: 0 - worse, max: 2 for Blocked and 12 for MEMI - better)
Time Frame: 1 week in each intervention condition
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Traumatic Brain Injury (TBI) Completing Intervention (MEMI Spaced Retrieval) | Non-Injured Comparison Participants Completing Intervention (MEMI Spaced Retrieval) | Participants With Traumatic Brain Injury (TBI) Completing Active Comparator (Blocked Retrieval) | Non-injured Comparison Participants Completing Active Comparator (Blocked Retrieval)
Number analyzed (Participants) | 19 | 20 | 19 | 20
units on a scale | 11.7 (0.6) | 11.8 (0.4) | 2 (0) | 2 (0)

3. Secondary Outcome: Free Recall of Word Forms
Description: Number of target word forms that participants type without cueing (0=did not remember any words- worse to 16=remembered all the words - better)
Time Frame: 1 week in each intervention condition
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Traumatic Brain Injury (TBI) Completing Intervention (MEMI Spaced Retrieval) | Non-Injured Comparison Participants Completing Intervention (MEMI Spaced Retrieval) | Participants With Traumatic Brain Injury (TBI) Completing Active Comparator (Blocked Retrieval) | Non-injured Comparison Participants Completing Active Comparator (Blocked Retrieval)
Number analyzed (Participants) | 19 | 20 | 19 | 20
score on a scale | 7.0 (3.4) | 10.9 (3.5) | 2.0 (2.9) | 4.0 (3.6)
Statistical Analysis 1: Comparison: Participants With Traumatic Brain Injury (TBI) Completing Intervention (MEMI Spaced Retrieval) vs Participants With Traumatic Brain Injury (TBI) Completing Active Comparator (Blocked Retrieval); Test type: Superiority — For preliminary efficacy, we used paired-samples t-tests within each group to compare free recall at the 1-week assessment between the two schedules; p < 0.001, t-test, 2 sided; degrees of freedom: 17; Mean Difference (Net) = 5.0 — Preliminary Intervention Effect = MEMI Free Recall - Blocked Free Recall
Statistical Analysis 2: Comparison: Non-Injured Comparison Participants Completing Intervention (MEMI Spaced Retrieval) vs Non-injured Comparison Participants Completing Active Comparator (Blocked Retrieval); Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.001, t-test, 2 sided; degrees of freedom: 19; Mean Difference (Net) = 6.8 — Preliminary Intervention Effect = MEMI Free Recall - Blocked Free Recall

4. Secondary Outcome: Cued Recall of Word Forms
Description: Number of target word forms that participants remember in response to prompting (i.e., typing the word that labels a given image) (0=did not remember any words- worse to 16=remembered all the words - better)
Time Frame: 1 week in each intervention condition
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Traumatic Brain Injury (TBI) Completing Intervention (MEMI Spaced Retrieval) | Non-Injured Comparison Participants Completing Intervention (MEMI Spaced Retrieval) | Participants With Traumatic Brain Injury (TBI) Completing Active Comparator (Blocked Retrieval) | Non-injured Comparison Participants Completing Active Comparator (Blocked Retrieval)
Number analyzed (Participants) | 19 | 20 | 19 | 20
score on a scale | 8.9 (5.0) | 12.1 (4.5) | 3.6 (3.4) | 6.8 (4.5)
Statistical Analysis 1: Comparison: Participants With Traumatic Brain Injury (TBI) Completing Intervention (MEMI Spaced Retrieval) vs Participants With Traumatic Brain Injury (TBI) Completing Active Comparator (Blocked Retrieval); Test type: Superiority — We used paired-samples t-tests within each group to compare cued word recall at the 1-week assessment between the two schedules; p < 0.001, t-test, 2 sided; degrees of freedom: 17; Mean Difference (Net) = 5.2 — Preliminary Intervention Effect = MEMI Cued Word Recall - Blocked Cued Word Recall
Statistical Analysis 2: Comparison: Non-Injured Comparison Participants Completing Intervention (MEMI Spaced Retrieval) vs Non-injured Comparison Participants Completing Active Comparator (Blocked Retrieval); Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, t-test, 2 sided; degrees of freedom: 19; Mean Difference (Net) = 5.3 — Preliminary Intervention Effect = MEMI Cued Word Recall - Blocked Cued Word Recall

5. Secondary Outcome: Cued Recall of Word Meanings
Description: Number of target word definitions that participants remember in response to prompting (i.e., typing the definition for a given word) (0=did not remember any words- worse to 16=remembered all the words - better)
Time Frame: 1 week in each intervention condition
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Traumatic Brain Injury (TBI) Completing Intervention (MEMI Spaced Retrieval) | Non-Injured Comparison Participants Completing Intervention (MEMI Spaced Retrieval) | Participants With Traumatic Brain Injury (TBI) Completing Active Comparator (Blocked Retrieval) | Non-injured Comparison Participants Completing Active Comparator (Blocked Retrieval)
Number analyzed (Participants) | 19 | 20 | 19 | 20
score on a scale | 11.3 (4.2) | 13.9 (3.0) | 7.7 (4.4) | 10.5 (4.6)
Statistical Analysis 1: Comparison: Participants With Traumatic Brain Injury (TBI) Completing Intervention (MEMI Spaced Retrieval) vs Participants With Traumatic Brain Injury (TBI) Completing Active Comparator (Blocked Retrieval); Test type: Superiority — We used paired-samples t-tests within each group to compare cued definition recall at the 1-week assessment between the two schedules; p = 0.003, t-test, 2 sided; degrees of freedom: 17; Mean Difference (Net) = 3.6 — Preliminary Intervention Effect = MEMI Cued Definition Recall - Blocked Cued Definition Recall
Statistical Analysis 2: Comparison: Non-Injured Comparison Participants Completing Intervention (MEMI Spaced Retrieval) vs Non-injured Comparison Participants Completing Active Comparator (Blocked Retrieval); Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.002, t-test, 2 sided; degrees of freedom: 19; Mean Difference (Net) = 3.3 — Preliminary Intervention Effect = MEMI Cued Definition Recall - Blocked Cued Definition Recall

6. Other Pre Specified Outcome: Number of Spatial Contexts
Description: At the beginning of each retrieval session, we ask participants to give their spatial context (the physical location in which they are completing the session, e.g., home or work). We report the number of different spatial contexts in which participants completed sessions in each condition. A higher number of spatial contexts indicates more variance in the contexts of retrieval opportunities, which is a goal of this technology (better).
Time Frame: 1 week in each intervention condition
Measure: Mean (Standard Deviation); unit: number of spatial contexts
Arm/Group | Participants With Traumatic Brain Injury (TBI) Completing Intervention (MEMI Spaced Retrieval) | Non-Injured Comparison Participants Completing Intervention (MEMI Spaced Retrieval) | Participants With Traumatic Brain Injury (TBI) Completing Active Comparator (Blocked Retrieval) | Non-injured Comparison Participants Completing Active Comparator (Blocked Retrieval)
Number analyzed (Participants) | 19 | 20 | 19 | 20
number of spatial contexts | 2.6 (1.4) | 2.9 (1.6) | 1.4 (0.5) | 1.2 (0.4)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Participants With Traumatic Brain Injury (TBI) Completing Intervention (MEMI Spaced Retrieval) | Non-Injured Comparison Participants Completing Intervention (MEMI Spaced Retrieval) | Participants With Traumatic Brain Injury (TBI) Completing Active Comparator (Blocked Retrieval) | Non-injured Comparison Participants Completing Active Comparator (Blocked Retrieval)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/19

LIMITATIONS AND CAVEATS:
Although participants were not incentivized for engagement, they were compensated for providing feedback on their experience. Participants may have been reluctant to provide critical feedback, but they were encouraged to provide their honest opinions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT06375421/Prot_001.pdf
  • Statistical Analysis Plan (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT06375421/SAP_002.pdf
  • Informed Consent Form (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT06375421/ICF_003.pdf